CLINICAL TRIAL: NCT02470390
Title: An Open-Label Single-Dose Crossover Study Comparing the Plasma and Cerebrospinal Fluid Pharmacokinetics and Bioavailability of Fentanyl Delivered Intranasally Versus Sublingually Versus Intravenously in Healthy Volunteers
Brief Title: Open Label Crossover Study Pharmacokinetics (PK) Study in Healthy Volunteers Receiving Various Forms of Fentanyl
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Depomed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: LAZA-PK-401
Record Dates: First submitted 2015-06-04; First posted 2015-06-12 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Volunteer; Pharmacokenetics (PK) (plasma and Cerebrospinal Fluid [CSF])
MeSH Terms: interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nasal fentanyl (Active Comparator): nasal fentanyl, 200 μg, administered as one 100 μg spray (100 μL) to each nostril; both completed within one minute.
  Will be administered on either study day 1 or 3 per protocol and randomization.
  Interventions: Drug: Fentanyl
- Sub-Lingual fentanyl (Active Comparator): sublingual fentanyl, 200 μg, administered as a single spray (100 μL) under the tongue.
  Will be administered on either study day 1 or 3 per protocol and randomization.
  Interventions: Drug: Fentanyl
- IV fentanyl (Active Comparator): IV fentanyl, 100 μg in 2 mL administered as an intravenous injection over 1-3 minutes.
  Will be administered on study day 5 per protocol.
  Interventions: Drug: Fentanyl

INTERVENTIONS:
Drug: Fentanyl — Lazanda (nasal spray), Subsys (sub-lingual) and intravenous fentanyl
  Other Names: Lazanda, Subsys, IV fentanyl

SUMMARY:
A partially randomized, open-label, 3-way crossover, single-center, systemic and CSF PK and bioavailability study in healthy volunteers.

DETAILED DESCRIPTION:
An Open-Label Single-Dose Crossover Study Comparing the Plasma and Cerebrospinal Fluid Pharmacokinetics and Bioavailability of Fentanyl Delivered Intranasally Versus Sublingually Versus Intravenously in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Normal healthy male or female between the ages of 18 to 65 years. Never smokers or Non-smokers (cessation of smoking ≥ 6 months ago). Body Mass Index (BMI = weight/height2) greater than or equal to 18.5 kg/m2 and less than or equal to 32.0 kg/m2.

No clinically meaningful findings in the physical examination, oral and nasal examination and 12-lead electrocardiogram.

Negative for drugs of abuse, alcohol, and nicotine. Negative for hepatitis A, B, and C and Human Immunodeficiency Virus (HIV). No clinical laboratory values outside of the acceptable range, unless, in the opinion of the Principal Investigator, they are deemed not clinically significant.

Exclusion Criteria:

* Subject has a known history of allergic reaction, hypersensitivity, or clinically significant intolerance to opioids, fentanyl or components of the study drugs.

  2. Subjects with a high potential for opioid addiction (personal or family history).

  3. Subject is lactating or considered at risk of pregnancy. 4. Subject has impaired liver function (e.g., alanine aminotransferase [ALT] ≥ 3 times the upper limit of normal [ULN] or bilirubin ≥ 3 times ULN), known active hepatic disease (e.g., hepatitis), or evidence of clinically significant liver disease or other condition affecting the liver that may suggest the potential for an increased susceptibility to hepatic toxicity with oral diclofenac exposure.

  5. Subject has any history of renal disease that, in the opinion of the investigator, would contraindicate study participation; or subject has significantly impaired renal function as evidenced by an estimated GFR of ≤60 ml/min/1.73m2.

  6. Subject has a history or evidence of significant nasal pathology, including polyps or nasal obstructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of R&D, Study Director — Depomed

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 13 healthy subjects were randomly assigned to treatment in this crossover study: 6 in the "Nasal Fentanyl First, then Sublingual Fentanyl and IV Fentanyl" arm and 7 in the "Sublingual Fentanyl First, then Nasal Fentanyl and IV Fentanyl" arm.
Groups:
- Nasal Fentanyl First, Then Sublingual Fentanyl and IV Fentanyl: Nasal Fentanyl, 200 μg, administered as one 100 μg spray (100 μL) to each nostril; both completed within one minute on Study Day 1 per protocol.
  Sublingual Fentanyl, 200 μg, administered as a single spray (100 μL) under the tongue on Study Day 3 per protocol.
  IV Fentanyl, 100 μg in 2 mL administered as an intravenous injection over 1-3 minutes on Study Day 5 per protocol.
- Sublingual Fentanyl First, Then Nasal Fentanyl and IV Fentanyl: Sublingual Fentanyl, 200 μg, administered as a single spray (100 μL) under the tongue on Study Day 1 per protocol.
  Nasal Fentanyl, 200 μg, administered as one 100 μg spray (100 μL) to each nostril; both completed within one minute on Study Day 3 per protocol.
  IV Fentanyl, 100 μg in 2 mL administered as an intravenous injection over 1-3 minutes on Study Day 5 per protocol.
Period: Overall Study
Arm/Group | Nasal Fentanyl First, Then Sublingual Fentanyl and IV Fentanyl | Sublingual Fentanyl First, Then Nasal Fentanyl and IV Fentanyl
Started | 6 | 7
Completed | 6 | 6
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Fentanyl First, Then Sublingual Fentanyl and IV Fentanyl | Sublingual Fentanyl First, Then Nasal Fentanyl and IV Fentanyl | Total
Number analyzed (Participants) | 6 | 7 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (14.38) | 43.0 (9.50) | 41.2 (11.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Fentanyl in Cerebrospinal Fluid (CSF) (1 of 3)
Time Frame: 6 hrs (pre-dose, 5, 10, 20, 30, 45, & 60 min, and 2, 3, 4, & 6 hrs post-dose on Study Days 1 & 3)
Population: The CSF PK population included all subjects who completed all study periods and Cmax was less than 5% pre-dose. The above CSF PK outcome compares nasal and sublingual fentanyl interventions.
Measure: Median (Full Range); unit: h
Groups:
- Nasal Fentanyl: Nasal Fentanyl, 200 μg, administered as one 100 μg spray (100 μL) to each nostril; both completed within one minute on Study Day 1 or 3 per protocol.
- Sublingual Fentanyl: Sublingual Fentanyl, 200 μg, administered as a single spray (100 μL) under the tongue on Study Day 1 or 3 per protocol.
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl
Number analyzed (Participants) | 10 | 9
h | 1.01 [0.75 to 3.00] | 2.00 [0.75 to 3.00]

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Fentanyl in Cerebrospinal Fluid (CSF) (2 of 3)
Time Frame: 6 hrs (pre-dose, 5, 10, 20, 30, 45, & 60 min, and 2, 3, 4, & 6 hrs post-dose on Study Days 1 & 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl
Number analyzed (Participants) | 10 | 9
pg/mL | 84.54 (47.10) | 56.37 (22.13)

3. Primary Outcome: Area Under the Concentration-Time Curve From Hour 0 to Hour 6 (AUC 0-6h) of Fentanyl in Cerebrospinal Fluid (CSF) (3 of 3)
Time Frame: 6 hrs (pre-dose, 5, 10, 20, 30, 45, & 60 min, and 2, 3, 4, & 6 hrs post-dose on Study Days 1 & 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg*h/mL
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl
Number analyzed (Participants) | 10 | 9
pg*h/mL | 300.25 (121.93) | 221.49 (76.82)

4. Primary Outcome: Maximum Observed Concentration (Cmax) of Fentanyl in Plasma (1 of 5)
Description: Cmax (pg/mL)
Time Frame: 24 hrs (pre-dose, 5, 10, 15, 20, 30, 45, & 60 min, and 1.5, 2, 3, 4, 6, 8, 12, & 24 hrs on Study Days 1 & 3 for Nasal Fentanyl / Sublingual Fentanyl; pre-dose, 2, 5, 10, 20, 30, & 60 min, and 2, 4, 6, 8, 12, & 24 hrs on Study Day 5 for IV Fentanyl)
Population: The Plasma PK population included all subjects who received at least 1 dose of study drug and had at least 1 evaluable PK parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Groups:
- IV Fentanyl: IV Fentanyl, 100 μg in 2 mL administered as an intravenous injection over 1-3 minutes on Study Day 5 per protocol.
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl | IV Fentanyl
Number analyzed (Participants) | 12 | 13 | 12
pg/mL | 541.28 (78.1) | 369.59 (41.4) | 1166.51 (130.8)

5. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 to the Last Quantifiable Concentration (AUC 0-tlast) of Fentanyl in Plasma (2 of 5)
Description: AUC 0-tlast (pg*h/mL)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl | IV Fentanyl
Number analyzed (Participants) | 12 | 13 | 12
pg*h/mL | 2752.51 (37.3) | 2359.08 (27.5) | 2236.46 (26.5)

6. Primary Outcome: Area Under the Concentration-Time Curve From Time 0 Extrapolated to Infinity (AUC 0-inf) of Fentanyl in Plasma (3 of 5)
Description: AUC 0-inf (pg*h/mL)
Time Frame: as for outcome 4
Population: The Plasma PK population included all subjects who received at least 1 dose of study drug and had at least 1 evaluable PK parameter. The AUC 0-inf values were excluded where %AUC extrap was greater than 20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl | IV Fentanyl
Number analyzed (Participants) | 6 | 7 | 3
pg*h/mL | 3413.80 (34.8) | 2879.85 (26.0) | 2871.89 (17.7)

7. Primary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Fentanyl in Plasma (4 of 5)
Description: Tmax (h)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: h
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl | IV Fentanyl
Number analyzed (Participants) | 12 | 13 | 12
h | 0.63 [0.17 to 2.00] | 0.75 [0.25 to 4.00] | 0.07 [0.03 to 1.00]

8. Primary Outcome: Terminal Elimination Half-Life (t1/2) of Fentanyl in Plasma (5 of 5)
Description: t1/2 (h)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl | IV Fentanyl
Number analyzed (Participants) | 10 | 12 | 6
h | 12.08 (40.0) | 10.73 (39.6) | 12.25 (24.2)

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Adverse Events were reported from the signed informed consent to 30 days after the last dose of study drug.
Arm/Group | Nasal Fentanyl | Sublingual Fentanyl | IV Fentanyl
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/13 | 0/12
Other Adverse Events (participants affected / at risk) | 2/12 | 6/13 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nasal Fentanyl (N=12) | Sublingual Fentanyl (N=13) | IV Fentanyl (N=12)
Post Lumbar Puncture Syndrome (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nasal Fentanyl (N=12) | Sublingual Fentanyl (N=13) | IV Fentanyl (N=12)
Nausea (Gastrointestinal disorders) | 1 | 3 | 0
Abdominal Distension (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Radicular Pain (Nervous system disorders) | 0 | 1 | 0
Catheter Site Pain (General disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees that sponsor shall have the right to the first publication of the study results which is intended to be a joint, multi-center publication. Following the first publication, the PI may publish study data or results, provided however PI submits the proposed publication to sponsor for review at least 60 days prior to the date of the proposed publication. Sponsor may remove any information that is considered confidential and / or proprietary other than study data.